CLINICAL TRIAL: NCT06350734
Title: Quality of Life After Treatment for Bladder Cancer: The Bladder Cancer Survivorship Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-004675; NCI-2024-00973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-004675 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-04-02; First posted 2024-04-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete surveys and also have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates the effect of bladder cancer treatment on quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare general and disease-specific quality of life outcomes at 6, 12, 24, and 36 months after treatment for localized bladder cancer using the PROMIS-29 and the Bladder Cancer Index (BCI) respectively.

II. To identify patient level characteristics that may influence quality of life outcomes after treatment for localized bladder cancer.

OUTLINE: This is an observational study.

Patients complete surveys and also have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed, clinically localized, bladder cancer
* Be willing to complete a survey in English before starting definitive treatment (surgery or radiation);
* Able to give consent.

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with clinically localized bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 704 (Estimated)
Dates: Start 2018-10-12 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life outcomes - PROMIS-29 | At baseline, 6, 12, 24, and 36 months
  Assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS)-29, a 29-item instrument with 29 questions in eight categories of Health Related Quality of Life (HRQOL): physical function, sleep disturbance, pain interference and pain intensity, fatigue, anxiety, depression) and ability to participate in social roles and activities. Questions are answered on a 5-point scale with varying responses assigned to the scale based on the category/question.
Change in quality of life outcomes - Bladder Cancer Index | At baseline, 6, 12, 24, and 36 months
  Assessed using the Bladder Cancer Index (BCI). The BCI consists of 36 items, with 4- or 5-point Likert response scales for each item, covering 3 primary domains: urinary (14 items), bowel (10 items), and sexual (12 items). The items focus on the frequency of the disease symptoms, with answer scales such as: "Never, rarely, about half the time, usually, or always".
Patient level characteristics | At baseline, 6, 12, 24, and 36 months after treatment
  Will be assessed by the effect of race/ethnicity, comorbid conditions, education level, gender, and age on patient reported outcomes. Interactions between intervention type and patient-level characteristics will be included. The distributions of variables will be summarized graphically and numerically.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Tyson, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials